CLINICAL TRIAL: NCT04481243
Title: Vaccine Effectiveness and Seroconversion to 23 Valent Pneumococcal Polysaccharide Vaccination in Children With Type 1 Diabetes
Brief Title: A Study to Evaluate Pneumococcal Polysaccharide Vaccine Effectiveness in Children With Type 1 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ana L. Creo, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 20-004356
Record Dates: First submitted 2020-07-20; First posted 2020-07-22 (Actual); Results first posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — 23-valent pneumococcal capsular polysaccharide vaccine; Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: Will study immunological response to vaccination
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pneumovax 23 (Experimental): Type 1 Diabetes subjects will receive Pneumovax 23-pneumococcal polysaccharide (PPSV23)
  Interventions: Biological: Pneumovax 23- pneumococcal polysaccharide; Procedure: Blood draw

INTERVENTIONS:
Biological: Pneumovax 23- pneumococcal polysaccharide — PPSV23 is a vaccine to help protect against serious infection due to the Streptococcus pneumoniae bacteria. One dose administered intramuscularly or subcutaneously.
  Other Names: PPSV23
Procedure: Blood draw — 6 ml blood draw at baseline and 6 months post immunization

SUMMARY:
The purpose of this study is to determine if children with type 1 diabetes have adequate immune response to PPSV23 vaccination and to assess factors affecting immune response.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 3-18 years old.
* Clinical diagnosis of Type 1 diabetes.

Exclusion Criteria:

* Newly diagnosed with Type 1 diabetes with in the past month of study date.
* Contraindications to receiving 23 valent pneumococcal vaccines.
* Other conditions associated with compromised immunity and vaccine response.
* Primary or Secondary Immune deficiency.
* Previous receipt of PPSV-23 vaccination.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Creo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ender E, Joshi A, Snyder M, Kumar S, Hentz R, Creo A. Seroconversion following PPSV23 vaccination in children with type 1 diabetes mellitus. Vaccine. 2025 Jan 25;45:126592. doi: 10.1016/j.vaccine.2024.126592. Epub 2024 Dec 11. PMID 39667114
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Pneumovax 23: Type 1 Diabetes subjects received Pneumovax 23-pneumococcal polysaccharide (PPSV23)
  Pneumovax 23- pneumococcal polysaccharide: PPSV23 is a vaccine to help protect against serious infection due to the Streptococcus pneumoniae bacteria. One dose administered intramuscularly or subcutaneously.
  Blood draw: 6 ml blood draw at baseline and 6 months post immunization
Period: Overall Study
Arm/Group | Pneumovax 23
Started | 29
Completed | 25
Not Completed | 4
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Pneumovax 23
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 11.6 (3.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 17
  Female | 11
  Unknown | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 27
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 28
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Immunoglobulin G (IgG) Antibodies
Description: Serological response. Blood draw for assessment of pneumococcal specific titer IgG. Measured as mcg/mL
Time Frame: 6 months post vaccination
Population: Three subjects withdrew prior to the 6 months post vaccination blood draw and one subject withdrew prior to receiving the vaccine.
Measure: Median (Inter-Quartile Range); unit: mcg/mL
Arm/Group | Pneumovax 23
Number analyzed (Participants) | 25
mcg/mL | 270.0 [203.3 to 270.1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study, approximately 6 months.
Arm/Group | Pneumovax 23
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-22): https://cdn.clinicaltrials.gov/large-docs/43/NCT04481243/Prot_SAP_000.pdf